CLINICAL TRIAL: NCT07295015
Title: Digital Maternal Support Tool Implementation: Research to Inform a Statewide Postpartum App Implementation Strategy
Brief Title: Digital Maternal Support Tool Implementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Tuscarora Intermediate Unit 11 (Unknown)
Responsible Party: Principal Investigator, Tamar Krishnamurti, Associate Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY24110002
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Postpartum
Keywords: postpartum; parenting; smartphone; mobile applications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postpartum support app (Experimental): All study participants will be given access to a postpartum support app. They will be asked to use this app for 8 weeks. Periodic surveys will be administered at 10 days, 4 weeks, and 8 weeks post enrollment. Baseline measurements will be collected at enrollment.
  Interventions: Other: Smartphone application

INTERVENTIONS:
Other: Smartphone application — The smartphone app is designed to provide postpartum education, screening and tracking, and positive parenting support for newly postpartum English-language speakers in Pennsylvania.

SUMMARY:
The goal of this trial is to learn if a smartphone app designed to provide postpartum support is acceptable to new mothers in Pennsylvania. The main questions it aims to answer are:

* How easy is the app is to use?
* Does the app meet the needs of new parents?
* Is using the app associated with better understanding of critical postpartum symptoms?
* Is using the app associated with endorsement of positive parenting statements?

Participants will:

* Use a postpartum support app on their smartphones for 8 weeks
* Answer survey questions about their experience

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the feasibility and acceptability of a smartphone app designed to provide postpartum education, screening and tracking, and positive parenting support for newly postpartum English-language speakers in Pennsylvania. This trial will also examine the preliminary effectiveness of the smartphone app for identifying symptoms and supporting positive parenting beliefs by measuring knowledge and attitude changes from pre-app use to post-app use.

ELIGIBILITY:
Inclusion Criteria:

* Recently delivered one or two live births at hospital recruitment site
* 18-45 years of age
* Can participate in English
* Has smartphone access for at least two months (study duration)

Exclusion Criteria:

* Did NOT recently deliver one or two live births at hospital recruitment site
* <18 or >45 years of age
* Cannot participate in English
* Does not have smartphone for at least two months (study duration)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of App | Day 10, Week 4, and Week 8 of study participation
  20 questions tailored from the Unified Theory of Acceptance of Use of Technology (UTAUT) asked at 3 study timepoints: 10 days, 4 weeks, and 8 weeks. 11 of the 20 questions are repeated across timepoints that assess the smartphone app (e.g., "The amount of information in [the app] is what I need" or "Overall, I like [the app]"). The remaining 9 are specific to distinct features of the app that are made available to the user at specific timepoints (e.g., "I like the way the healing check-in looks and feels"; "I like the way the [2-month] baby milestones look and feel"). Answers are measured on a 5-point Likert scale, ranging from (1)strongly disagree to (5) strongly agree (5), unless reverse-coded. Means and standard deviations will be calculated for each item, with higher responses indicating higher levels of acceptability.
Feasibility of App Use | From enrollment (baseline) to the end of study participation at 8 weeks.
  Feasibility will be measured using rate of engagement. Engagement will be evaluated by the number of study weeks that users uniquely access the smartphone app.

SECONDARY OUTCOMES:
Knowledge - postpartum symptoms | Enrollment (baseline), day 10, week 4, and week 8 of study participation
  From a list of 14 postpartum symptoms, participants will be asked to classify the symptom with the appropriate response: monitor at home, call your provider, or call 911/seek emergency care. Baseline knowledge will be measured at enrollment based on the number correct out of 14, with follow-up measurements taken at 10 days, 4 weeks, and 8 weeks.
Attitudes - positive parenting | Enrollment (baseline), day 10, week 4, and week 8 of study participation
  From a list of 10 statements focused on parenting practices, participants will rate the statements from strongly disagree (1) to strongly agree (5). Example statements include, "Skin-to-skin contact improves baby health and development," "Babies need strict routines" (reverse coded), and "Infants should be fed when they show hunger cues." These responses are summed, with higher scores indicating stronger endorsement of positive parenting. These measurements are taken as a baseline measurement at enrollment, and then again at 10 days, 4 weeks, and 8 weeks.

OTHER OUTCOMES:
Health services utilization | Day 10, week 4, and week 8 of study participation
  Well-visit (maternal) and check-up (infants) attendance are surveyed on day 10, week 4, and week 8 (e.g., "Has your baby (or twins) had their first well visit with their pediatrician yet?" or "Have you attended a postpartum check-up?"). Non-routine healthcare utilization is surveyed at week 4 and week 8 (e.g., "In the last 4 weeks, did your baby (or twins) have a visit at an emergency department?"or "In the last 8 weeks, did you call, message or schedule a visit with your Obstetrician or Primary Care Provider for a reason other than a postpartum check-up?"). Distributions for each response will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Krishnamurti, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://myana-app.com